CLINICAL TRIAL: NCT04412005
Title: Pregnant Women as a Sentinel Group for Malaria Surveillance in an Era of Changing Malaria Transmission
Brief Title: Pregnant Women for Malaria Surveillance
Acronym: MiPMon
Status: Completed | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01AI123050 (NIH)
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: P. Falciparum
Keywords: malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots Plasma and PBMCS from a random selection of study participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Manhiça: Pregnant women attending the Manhiça District Hospital
  Interventions: Other: No intervention
- Ilha Josina: Pregnant women attending the Ilha Josina Health Center
  Interventions: Other: No intervention
- Magude: Pregnant women attending the Magude Health Center
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Close monitoring of malaria in pregnancy can help to quickly identify changes in malaria burden and related adverse outcomes, especially in areas embarking in malaria elimination activities. The easy access of pregnant women through antenatal clinics, combined with the potential of pregnancy-specific serology to assess cumulative exposure to malaria, can provide the basis for new sentinel surveillance methods. Such an approach has the potential to guide clinical practice and the choice of malaria control/preventive tools adapted to areas of different transmission intensity, as well as to generate sensitive metrics of transmission during malaria elimination activities.

DETAILED DESCRIPTION:
Continued monitoring of malaria in pregnancy is lacking in most endemic settings, in spite of its significant disease burden. Increases in malaria-related harmful effects observed among Mozambican pregnant women after drastic malaria declines during the last decade [2] suggest that closely monitoring of the transmission is needed to quickly identify rebounds in adverse outcomes, especially in areas embarking in malaria elimination activities. Moreover, several evidences point to IgGs against VAR2CSA (the parasite antigen that mediates sequestration of P. falciparum in the placenta) as a marker of cumulative exposure to P. falciparum during pregnancy that can provide estimates of malaria transmission. The investigators hypothesize that dynamics of malaria in pregnancy and pregnancy-specific immunity reflect changes in the intensity of transmission through location and time, not only among pregnant women but also in the underlying community. The goal of this study is to provide epidemiological, molecular and immunological insights of the value of pregnant women attending health facilities to generate estimates of malaria burden and its adverse consequences in situation of varying levels of malaria transmission, with the ultimate hope of developing new tools for the monitoring of malaria in endemic countries. To address this, the investigators will conduct a three-year prospective observational study at three health facilities with different levels of malaria transmission in Maputo Province to determine the relationship between malaria transmission, parasitological outcomes and the clinical impact of malaria infection in pregnant women at their first antenatal visit, delivery and during sick visits (Aim 1.1). Moreover, the investigators will create a sample repository biobank for future investigations on host and parasite factors influencing malaria disease during pregnancy (Aim 1.2). The investigators will also determine the relationship between malaria estimates obtained from pregnant women, children at hospital visits, (Aim 2.1) and seroprevalences against VAR2CSA (Aim 2.2). The impact of interrupting malaria transmission on pregnancy-specific serology (Aim 2.3) will be assessed in pregnant women from Magude after mass drug administration in the community. Finally, scientific capacity in the Manhiça Health Research Center (Aim 3) will be developed through training on a) epidemiological research and management of malaria data; b) molecular tools for detection of malaria parasites and molecular markers of antimalarial resistance for rapid mapping of drug resistance; and c) pregnancy-specific immunity as an innovative tool to assess malaria transmission. This study will contribute to promote a pregnancy malaria research agenda by improving our scientific knowledge on determinants of malaria susceptibility during pregnancy and demonstrating the feasibility and value of an easy-to-implement new generation serological tool for malaria surveillance in malaria elimination contexts.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending their first routine ANCs or pregnant women seen at the moment of delivery or pregnant women with signs/symptoms of malaria (axillary temperature ≥ 37.5°C, referred history of fever in the last 24 hours, pallor, arthromyalgias, headache and/or history of convulsions)
* Being equal or older than 16 years
* Being from the study area

Exclusion Criteria:

* Unwillingness to participate in the study or to have samples obtained
* Not being from the study area.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Being pregnant
Study Population: Pregnant women attending three health centers in areas of Maputo Province with different levels of malaria transmission (Manhiça District Hospital [Manhiça District], Ilha Josina Health Center [Manhiça District] and Magude Health Center [Magude District])
Sampling Method: Non-Probability Sample
Enrollment: 16958 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Number of pregnant women with a P. falciparum infection | 3 years
  P. falciparum detected by qPCR

SECONDARY OUTCOMES:
Number of pregnant women with maternal anemia | 3 years
  Hemoglobin levels (Hemocue)
Number of pregnant women delivering a newborn with low birthweight | 3 years
  grams in a digital scale

IPD SHARING:
Plan to Share IPD: Undecided